CLINICAL TRIAL: NCT02842567
Title: Hydroxytyrosol and Vitamin E in the Treatment of Children With Biopsy-proven NASH
Brief Title: Hydroxytyrosol and Vitamin E in Pediatric NASH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Valerio Nobili, Professor, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1066_OPBG_2016
Record Dates: First submitted 2016-07-13; First posted 2016-07-25 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2017-07

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 3,4-dihydroxyphenylethanol; Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATED GROUP (Experimental): This group will treated with 2 pills daily, each containing 3.75 mg of hydroxytyrosol plus 5 mg of Vitamin E, given orally for 16 weeks.
  Interventions: Drug: Hydroxytyrosol plus Vitamin E
- PLACEBO GROUP (Placebo Comparator): This group will treated with 2 identical placebo pills daily given orally for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxytyrosol plus Vitamin E — This group will treated with 2 pills daily, each containing 3.75 mg of hydroxytyrosol plus 5 mg of Vitamin E, given orally for 16 weeks
  Other Names: Hydroxytyrosol, alpha-tocopherol
  Arms: TREATED GROUP
Drug: Placebo — This group will treated with 2 identical placebo pills daily given orally for 16 weeks.
  Arms: PLACEBO GROUP

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) has reached epidemic proportions and is rapidly becoming the one of most common causes of chronic liver disease in children. The pathogenesis of NAFLD is generally considered the result of a series of liver injuries, commonly referred as "multi-hit" hypothesis. Several studies suggest that inflammatory pathways and oxidative stress could be responsible of disease progression to non-alcoholic steatohepatitis (NASH).

Hydroxytyrosol is a simple phenolic compound naturally occurring in olive and olive oil with antioxidant properties. Some studies have demonstrated that hydroxytyrosol show several anti-inflammatory and anti-atherogenic activities, such as the inhibition of LDL oxidation and platelet aggregation.

Alpha tocopherol (Vitamin E) is the most studied anti-oxydant in pediatric NAFLD with conflicting results. It inhibits proinflammatory cytokine production and attenuates the release of profibrogenic agents and liver collagen.

The purpose of this interventional study is to evaluate the efficacy and tolerability of Hydroxytyrosol and Vitamin E in the treatment of children with biopsy-proven NASH.

DETAILED DESCRIPTION:
80 children and adolescents (4-16 years) with biopsy-proven NASH will be enrolled. They will be randomized to treatment with hydroxytyrosol and vitamin E (n: 40 pts) or an identical placebo (n: 40 pts) given orally for a period of 16 weeks. Patients will undergo a medical evaluation at baseline (enrollment) and after 4 months (end of treatment). Anthropometric measures and laboratory assay, includin liver enzymes, gluco-insulinemic and lipid profiles will be performed at baseline and at the end of the study. Hepatic ultrasound examination will be performed at enrollment and at the end of the study.

Serum sample for determination of markers of inflammation and oxidative stress will be collected at enrollment and at the end of the study.

A stool sample for analysis of gut microbioma will be collected at enrollment and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy consistent with diagnosis of NASH (liver biopsy performed in 3-6 months before enrollment)
* Hyperechogenicity of liver at ultrasound examination
* ALT levels range between normal and < 10 UNL
* INR < 1.3
* Albumin > 3 gr/dl.
* Total bilirubin < 2.5 mg/dl
* normal renal function
* normal cells blood count
* exclusion of other causes of chronic hepatopathies in children
* Written informed consent to participate in the Protocol by their parents or legal guardians of patients

Exclusion Criteria:

* alcohols or drugs abuse
* use of drugs known to induce steatosis or to affect body weight or carbohydrate metabolism
* autoimmune liver diseases, Wilson's disease, alpha-1-antitripsin deficiency, metabolic liver disease
* every clinical or psychiatric diseases interfering with experimentation according to investigator's evaluation
* finding of active liver disease due to other causes

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Improvement of laboratory markers of inflammation and oxidative stress, such as concentrations of TNF-alpha, lipopolysaccharide (LPS), adiponectin, catepsin D, cytokeratin-18. | 4 months
Improvement of laboratory parameters of metabolic syndrome, such as lipids and gluco-insulinemic profile, transaminases serum levels | 4 months

SECONDARY OUTCOMES:
Improvement of echographic score of hepatic steatosis (echographic scale) | 4 months
Number of participants with treatment-related adverse events as assessed by CTCAE | 4 months
Analysis of fecal gut microbiome of patients before and after treatment with hydroxytyrosol and vitamin E | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatometabolic Department, Bambino Gesù Children's Hospital, Rome, Italy

REFERENCES:
- [Derived] Mosca A, Crudele A, Smeriglio A, Braghini MR, Panera N, Comparcola D, Alterio A, Sartorelli MR, Tozzi G, Raponi M, Trombetta D, Alisi A. Antioxidant activity of Hydroxytyrosol and Vitamin E reduces systemic inflammation in children with paediatric NAFLD. Dig Liver Dis. 2021 Sep;53(9):1154-1158. doi: 10.1016/j.dld.2020.09.021. Epub 2020 Oct 13. PMID 33060043